CLINICAL TRIAL: NCT03186885
Title: Healthy Frio: A Rural Community Partnership to Advance Latino Obesity Research
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Texas at Austin (Other)
Collaborators: The University of Texas at San Antonio (Other); The University of Texas Health Science Center at San Antonio (Other); University of Maryland (Other)
Responsible Party: Principal Investigator, Deborah Parra-Medina, Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01NR016269 (NIH)
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Obesity; Nutrition Poor; Physical Activity; Weight Loss
MeSH Terms: conditions — Obesity; Malnutrition; Motor Activity; Weight Loss

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- In-Person Family Intervention (Experimental): Healthy Frio In-Person Family-focused Intervention; In-person group setting at a community center
  Interventions: Behavioral: Healthy Frio In-Person Family-focused Intervention
- Remote Technology Family Intervention (Experimental): Healthy Frio Remote Technology Family-focused Intervention; Home-based delivered remotely with technology
  Interventions: Behavioral: Healthy Frio Remote Technology Family-focused Intervention
- Control (Active Comparator): Control; Participants will receive standard health education materials, a community resource guide, and encouragement to follow up with their primary care provider for office-based counseling.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Healthy Frio In-Person Family-focused Intervention — Participants learn about energy balance behaviors, skills to support health behavior change, managing personal wellness, and parenting strategies. Sessions use interactive learning strategies to elicit knowledge and experience of participating families to encourage families to learn from each other. YMCA staff members lead a 50-minute group exercise session after each health education session to help participants meet their commitment of engaging in PA at least 3 times/week.
  Other Names: FI-IP
  Arms: In-Person Family Intervention
Behavioral: Healthy Frio Remote Technology Family-focused Intervention — Tablet computers will be used as the platform to deliver the health education content for the FI-RT. Each session will present the class content and guide the participants to complete class activities. Videos of health education and class activities (e.g., cooking demonstrations, exercise demonstrations) will be embedded in the lesson. Interactive assessment questions with feedback will be presented throughout the session to check for understanding of the content. Viewing time and responses to the assessment questions will be recorded to evaluate progress and comprehension. Participants will view the health education sessions at home as a family and discuss the content as prompted by lesson instructions.
  Other Names: FI-RT
  Arms: Remote Technology Family Intervention
Behavioral: Control — Participants receive standard of care
  Arms: Control

SUMMARY:
Much has been learned about the efficacy and effectiveness of comprehensive healthy lifestyle interventions to reduce obesity. Few studies have been translated into rural settings or among Latinos. Y Living is an evidence-based family-focused intervention (FI) designed for urban Latino families. The FI is a 12-week behavioral modification program grounded in social cognitive theory, designed to engage the whole family in lifestyle changes by developing knowledge and skills in physical activity and healthy eating, building skills in goal-setting and self-monitoring, and creating a supportive home environment. Researchers will engage community partners in formative research to adapt the current FI for rural Latino families. Two parallel delivery methods of the FI will be developed and tested: 1) in-person group setting at a community center (FI-IP) and 2) home-based delivered remotely with technology (FI-RT). Both will be designed to address the unique social, cultural and environmental factors facing rural Latino families. The FI-RT will take advantage of innovative modern technology and e-Learning to increase program availability, accessibility and participation in rural settings. Researchers will conduct a 3-arm randomized controlled trial (RCT) to compare effectiveness of the two delivery approaches on weight loss (primary outcome) and energy balance behaviors (secondary outcomes) among obese Latino parent-child pairs versus control. The researchers will recruit 270 obese Latino adults (ages 21-65) with a child (ages 8-17) from three primary care practices in rural South Texas. These parent-child pairs will be randomized to one of three arms stratified by clinic: 1) FI-IP (n=90); 2) FI-RT (n=90); or 3) control group (n=90). Primary specific aims are to: 1) Conduct community-engaged formative studies to transform the existing FI into two unique delivery methods (FI-IP and FI-RT) for use in a subsequent RCT in a rural Latino community; and 2) Conduct a RCT to evaluate the comparative effectiveness of FI-IP and FI-RT to address weight loss (primary outcome) and energy balance behaviors (secondary outcomes) among obese rural Latino adults compared with adult participants in control group at immediate post intervention (3 months), after a 3-month maintenance program (6 months post randomization) and a 6-month follow-up (12 months post randomization). A secondary aim is to examine the impact of FI-IP and FI-RT children's weight and energy balance behaviors.

DETAILED DESCRIPTION:
Obesity is a significant health threat in South Texas, a largely Latino region with one of the most underserved, at-risk populations in the nation. Obesity can start in early childhood and persist lifelong, setting the stage for disease.1-3 Because obesity impairs health-related quality of life and billions are spent to manage obesity-related diseases,4 interventions to help obesity-affected families to adopt and maintain a healthier lifestyle and achieve a healthy weight can have great individual and public health benefits.

Much has been learned about the efficacy and effectiveness of comprehensive healthy lifestyle interventions to reduce obesity, but few studies have been translated into rural settings or for Latinos.5 Barriers to implementing lifestyle interventions in rural settings include: limited accessibility to health promotion programs, lack of health infrastructure, transportation constraints, poverty, and low levels of health literacy.6,7 To address these challenges, the proposed study will test two different methods of delivering a family-focused, culturally appropriate healthy lifestyle intervention to obese Latino adults and their families in rural South Texas. The family-focused intervention (FI), which builds on evidence from studies of urban Latino families by PI Dr. Deborah Parra-Medina and her South Texas-based research team, is a 12-week behavioral modification program grounded in the social cognitive theory of behavior change. The intervention is designed to engage the whole family in lifestyle changes by developing knowledge and skills in physical activity (PA) and healthy eating, building skills in goal-setting and self-monitoring, and creating a supportive environment at home.

Two parallel delivery methods of the FI will be developed and tested: 1) in-person group setting at a community center (FI-IP) and 2) home-based delivered remotely with technology (FI-RT). While both will be designed to address the unique social, cultural and environmental factors facing rural Latino families, the latter takes advantage of innovative technology and e-Learning to increase program availability, accessibility and program participation in rural settings. The investigators will conduct a 3-arm randomized controlled trial to compare the effectiveness of the two delivery approaches on weight loss (primary outcome) and energy balance behaviors (secondary outcomes) among obese Latino parent-child pairs versus control. The investigators will recruit 270 obese (BMI 30-39.9kg/m2) Latino adults (ages 21-65) with a child (ages 8-17) from three primary care practices in rural South Texas. These 270 parent-child pairs will be randomized to one of three arms stratified by clinic: 1) FI-IP (n=90); 2) FI-RT (n=90); or 3) control group (n=90). The primary specific aims of the study are:

Aim 1: Conduct community-engaged formative studies to transform the existing family-focused intervention (FI) into two unique delivery methods (FI-IP and FI-RT) for use in a subsequent randomized controlled trial in a rural Latino community.

Aim 2: Conduct a randomized controlled trial to evaluate the comparative effectiveness of two parallel delivery methods of family-focused intervention (FI-IP and FI-RT) to address weight loss (primary outcome) and energy balance behaviors (secondary outcomes) among obese rural Latino adults compared with control group adults at immediate post intervention (3 months post randomization), again after a 3-month maintenance program (6 months post randomization) and a 6-month follow-up (12 months post randomization).

• The investigators hypothesize that adult participants randomized to either FI-IP or FI-RT will achieve greater weight loss and improved energy balance behaviors compared with adult participants in the control group immediate post intervention (3 months post randomization), after a 3-month maintenance program (6 months post randomization) and a 6-month follow-up (12 months post randomization).

The secondary aims are to examine:

* the impact of family-focused interventions on children's weight and energy balance behaviors;
* the impact of the family-focused interventions on health-related quality of life (HRQOL);8 and
* factors that facilitate or impede implementation and adherence to the two intervention forms.

Findings from this comparative effective research will contribute to the evidence base to inform clinical and health policy decisions in regard to weight management for obese patients who may benefit from different approaches in intervention delivery.9 If successful, the remote delivery approach holds great promise in improving healthcare to underserved populations in rural and other remote locales.

ELIGIBILITY:
Inclusion Criteria:

* The investigators will recruit persons (index parent) who meet the following criteria: a) self-identified Latino adult; b) overweight or obese (BMI >= 25 kg/m2); c)not currently enrolled in a formal weight loss program or taking weight loss medications; d) no restriction for PA (i.e., no significant physical disability); e) having a smart phone;f) speaks and reads English; g) one child aged 8-17 (with no regard to obesity status) residing with the parent full-time and willing to participate; and h) receiving care at a study clinic.

Exclusion Criteria:

* Has a physical disability restricting physical activity
* Has a cognitive impairment

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Weight | Baseline, 3 months, 6 months 12 months
  Measured (to the nearest 0.1 kg.
Change in Percent body fat | Baseline, 3 months, 6 months 12 months
  Measured by bioelectrical impedance analysis (BIA) using the foot-to-foot pressure contact electrode BIA technique using a portable Tanita Body Composition Analyzer following standard protocol.
Change in Waist circumference (minimum waist girth) | Baseline, 3 months, 6 months 12 months
  Will be measured to the nearest 0.1 cm using a retractable, tension-controlled metal tape measure at the midway between the right iliac crests and the lower ribs when the subject is standing erect with feet together.
Change in BMI | Baseline, 3 months, 6 months 12 months
  BMI will be calculated as weight (kg)/height squared (m2) for adults and BMI percentile for age and gender for children.

SECONDARY OUTCOMES:
Physical Activity (objective) | Baseline, 3 months, 6 months 12 months
  Parent and child PA level will be assessed using the Actigraph (Fort Walton Beach, FL) accelerometers worn for 7 consecutive days recording 15-second epochs. Participants must wear the accelerometer for at least 12 hours per day and on at least 4, including on weekend day, of the 7 days for reliable measurement of activity. Total minutes per day in Moderate-to-vigorous physical activity and sedentary activity will be computed with MeterPlus Software Version 4.3.
Physical Activity (self-report) | Baseline, 3 months, 6 months 12 months
  To characterize participants' type, pattern, nature, and amount of PA, a comprehensive self-report measure will be administered, the Block Energy Expenditure Survey for adults, which measures total average energy expenditure per day and minutes per day of moderate and vigorous activities by activity type. For children, we will use the Block Kids Physical Activity Screener for school-age children and adolescents. It asks about frequency and duration of activities in the past 7 days with 9 items about leisure and school activities, chores and part-time jobs. It also asks about sedentary behavior (time spent with TV, video games, and Internet).
Dietary Intake | Baseline, 3 months, 6 months 12 months
  We will use a validated Block Food Frequency Questionnaire (FFQ) for adults and children (2005 FFQ for Adults and 2004 FFQ for Kids ages 8-17). The correlation between the FFQ and 24-hr recalls for energy intake (0.5) and nutrients (≥ 0.4) are satisfactory. FFQ is interviewer-administered by trained bilingual research staff using a visual portion-size graphic to facilitate accurate estimation of quantities consumed. This questionnaire estimates usual and customary intake of a wide array of nutrients and food groups with additional food items typical of diets among Latinos.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Parra-Medina, PhD, Principal Investigator — The University of Texas at Austin
Locations (1):
- South Texas Rural Health Services Clinic, Pearsall, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yin Z, Errisuriz VL, Evans M, Inupakutika D, Kaghyan S, Li S, Esparza L, Akopian D, Parra-Medina D. A Digital Health Intervention for Weight Management for Latino Families Living in Rural Communities: Perspectives and Lessons Learned During Development. JMIR Form Res. 2020 Aug 20;4(8):e20679. doi: 10.2196/20679. PMID 32726748
- See also: A Digiral Health Intervention for Weight Management For Latino Families Living in Rural Communities — http://formative.jmir.org/2020/8/e20679/